CLINICAL TRIAL: NCT03485495
Title: Multicenter Double-blind Placebo-controlled Randomized Parallel-group Clinical Study of Efficacy and Safety of Divaza for Adjustment of Oxidative Disorders in Patients With Cerebral Atherosclerosis
Brief Title: Clinical Trial of Efficacy and Safety of Divaza for Adjustment of Oxidative Disorders in Patients With Cerebral Atherosclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-DV-010
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis | interventions — divaza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Divaza (Experimental): Tablet for oral use. Two tablets per intake 3 times a day (approximately at the same time), outside of meal (between meals or 15 minutes before eating or drinking). The tablets should be held in mouth until completely dissolved.
  Interventions: Drug: Divaza
- Placebo (Placebo Comparator): Tablet for oral use. Two tablets per intake 3 times a day (approximately at the same time), outside of meal (between meals or 15 minutes before eating or drinking). The tablets should be held in mouth until completely dissolved.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Divaza — Oral administration.
  Arms: Divaza
Drug: Placebo — Oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to obtain additional data on efficacy and safety of Divaza for adjustment of oxidative disorders in patients with cerebral atherosclerosis.

It is assumed that the inclusion of the drug Divaza in the basic therapy will help reduce the severity of cognitive disorders, other clinical symptoms of cerebral atherosclerosis, reduce the impact of the disease on the quality of life of the patient.

Participate in the study may be patients with a diagnosis of "cerebral atherosclerosis", which, against the backdrop of basic therapy with constant doses of drugs (within the last 4 weeks), to achieve a stable course of cerebral atherosclerosis, cognitive disorders without significant disability are detected.

DETAILED DESCRIPTION:
Design - a multicenter randomized double-blind placebo-controlled parallel-group clinical trial.

The study will enroll the patients of either gender aged 40-75 years old inclusively with verified atherosclerotic cerebrovascular lesions (ICD-10 code - "Cerebral atherosclerosis" [I67.2]), with cognitive disorders (МоСА<26), without relevant incapacity (mRs≤1).

At screening visit (Visit 1, from day - 5 to day 0), after signing patient information sheet (informed consent form) for participation in the clinical study the patient's complaints and medical history will be collected and objective examination will be carried out. The investigator will assess intensity of cognitive disorders using MoCA, extent of functional capacity using mRs .

If the patient meets inclusion criteria and has no exclusion criteria at Visit 2 (Day 0) he/she will be randomized to one of two groups: group 1 will receive Divaza at 2 tablets 3 times a day; group 2 - placebo using study drug scheme.

Laboratory examination will be performed.

1. oxidant and antioxidant systems (Fe2+-induced chemoluminescence method, ELISA) defining: 1.1. level of preformed LP products, predominantly lipid hydroperoxides; 1.2. low and very low density lipoprotein resistance to LP; 1.3. lipoprotein potential for oxidation; 1.4. serum NO product concentration (Griess reaction).
2. compensatory potential of endothelium and its ability for adequate regulation of vascular tone with : 2.1. determination of platelet aggregation with bandage sign; 2.2. MAH duplex scanning. Procedures of Visit 2 may be performed on day of Visit 1 if general rules for blood collection are met, at that previously performed procedures will not be repeated.

The first administration of Divaza or Placebo will be performed at Visit 2 at medical site in the investigator's presence. The patient monitoring and therapy will last for 12 weeks during which 3 additional visits will be made.

At Visit 3 (Week 4±5 days) the investigator will collect the complaints, perform objective examination, evaluate intensity of cognitive disorders (MoCA). The investigator will monitor the prescribed, basic and concomitant therapy, evaluate therapeutic safety.

At Visit 4 (Week 8±5 days) the investigator will make a phone call to the patient to evaluate safety of the treatment.

At the final Visit 5 (Weeks 12±5 days) the investigator will evaluate intensity of cognitive disorders (MoCA). Laboratory examination of oxidant and antioxidant systems, compensatory potential of endothelium and its potential for adequate vascular tone regulation. The investigator will monitor the prescribe, basic and concomitant therapy, evaluate therapeutic safety and treatment compliance.

During the study basic, concomitant therapy will be allowed except for the products indicated in the section "Prohibited concomitant therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders aged 40-75 years old inclusive.
2. Diagnosis of cerebral atherosclerosis verified by all three signs:

   * underlying vascular disease (atherosclerosis and/or hypertension) and focal neurological symptoms combined with cerebral symptoms (headache, dizziness, tinnitus, impaired memory, working capacity);
   * ultrasound signs of atherosclerotic cerebrovascular lesions (according to MAH duplex scanning within 6 months preceding the patient enrollment into the study);
   * signs of morphological changes in the brain based on neuroimaging (CT/MRI 1.0-1.5 T) (subcortical and periventricular leukoaraiosis and/or focal changes in grey matter and white matter in the form of postischemic cysts and/or lacunar strokes and/or diffuse atrophic changes in the form of dilated cardiovascular system or subarachnoidal spaces).
3. Cognitive disorders (MoCa <26).
4. Patients with unchanged dose and combination of basic therapy of cerebral atherosclerosis and hypertension during the previous month.
5. Patients who gave their consent to use reliable contraception during the study.
6. Availability of signed patient information sheet and informed consent form for participation in the clinical trial.

Exclusion Criteria:

1. History of subarachnoidal/parenchymatous/ventricular hemorrhage, cerebral tumour or another disease resulting in neurological disorders.
2. Ischemic-type stroke or any other acute cerebrovascular accident less than 6 months prior to the study with Modified Rankin Scale (mRs) > 1 .
3. Cardiac sources of high risk or medium risk embolism (TOAST criteria).
4. Signs of acute or exacerbated chronic infectious diseases at or less than 2 weeks prior to screening.
5. History of CNS diseases including:

   * Inflammatory CNS diseases (G00-G09)
   * Systemic Atrophies Primarily Affecting the CNS (G10-G13)
   * Other degenerative diseases of the nervous system (G30-G32)
   * Demyelinating diseases of the CNS (G35-G37).
6. Dementia (F00-F03).
7. Previously diagnosed cardiovascular diseases with functional class III or IV (according to New York Heart Association, 1964).
8. Hypothyroidism, diabetes mellitus and other somatic diseases at decompensation stage.
9. Uncontrollable hypertension: SBP > 180 mm Hg and/or DBP > 110 mm Hg.
10. Diseases of lower limb veins (lower limb varicose veins, deep venous thrombosis, etc.) at decompensation stage.
11. Any other severe concomitant pathology which, according to the investigator, may interfere with the patient's participation in the study.
12. History/suspicion of oncology of any location (except for benign neoplasms).
13. Allergy/intolerance of any component of the drug products used in the therapy.
14. Hereditary lactose intolerance.
15. Malabsorption syndrome, including congenital or acquired lactase deficiency (or any other disaccharidase deficiency) and galactosemia.
16. Pregnancy, breast-feeding.
17. History of treatment non-compliance, psychiatric disorders, alcoholism or drug abuse which, according to the investigator, may interfere with the study procedures.
18. Use of any medicine indicated in the section "Prohibited concomitant treatment" within 1 month prior to enrollment.
19. Participation in other clinical trials in the previous 3 months.
20. Patients who are related to any of the on-site research personnel directly involved in the study or are an immediate relative of the study investigator, or has another conflict of interests. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
21. Patients who work for OOO "NPF "MATERIA MEDICA HOLDING" (i.e. the company's employees, temporary contract workers, appointed officials responsible for carrying out the research or immediate relatives of the aforementioned).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - Limited Liability Company "Family policlinic no. 4", Korolyov
  - Moscow City Clinical Hospital after V.M. Buyanov, Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow City Clinical Hospital No. 1 named after. N.I. Pirogov Moscow Department of Health, Moscow
  - Federal State Budgetary Institution Federal Research and Clinical Center of Physical-Chemical Medicine Federal Medical Biological Agency, Moscow
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Budget Scientific Institution "Scientific Center of Neurology", Moscow
  - The state budgetary health care institution of the Vladimir region "Regional Clinical Hospital", Vladimir
  - Federal State Budgetary Educational Institution of Higher Education "Yaroslavl State Medical University" of the Ministry of Healthcare of the Russian Federation, Yaroslavl
  - State Institution of Health of the Yaroslavl Region Clinical Hospital No. 8, Yaroslavl
  - State budgetary institution of health care of the Yaroslavl region "Regional Clinical Hospital", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Divaza | Placebo
Started | 65 | 59
Completed | 64 | 59
Not Completed | 1 | 0
Not completed — Non-compliance with inclusion criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Divaza | Placebo | Total
Number analyzed (Participants) | 65 | 59 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (7.8) | 59.8 (7.4) | 60.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 40 | 91
  Male | 14 | 19 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 65 | 59 | 124

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Value of Lipoprotein Resistance to LPO.
Description: Based on laboratory evaluation. Change in the mean resistance of lipoprotein (LP) to lipid peroxidation (LPO) after 12-week therapy versus baseline.
Time Frame: 12 weeks of the observation period.
Population: 1 patient in Divaza group had no laboratory data.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Divaza | Placebo
Number analyzed (Participants) | 63 | 59
seconds
  Resistance of LP to LPO at baseline | 42.4 (13.1) | 42.9 (11.2)
  Resistance of LP to LPO after 12 weeks | 55.6 (12.5) | 49.4 (14.3)
  ∆ between baseline and after 12 weeks | 14.8 (14.7) | 6.4 (16.9)
Statistical Analysis 1: Comparison: Divaza vs Placebo; This analysis applies to ∆ between baseline and after 12 weeks row; Test type: Superiority; p = 0.007, t-test, 2 sided — A priori threshold for statistical significance is split evenly between primary and secondary endpoints. α=0.025

2. Secondary Outcome: Percentage of Patients With Improved Cognitive Function.
Description: MoCA (Montreal Cognitive Assessment) score +1 and over after 12-week therapy versus baseline. Minimum score is 0, maximum score is 30. Higher values represent a better outcome.
Time Frame: 12 weeks of the observation period.
Population: 8 patients in Divaza group and 2 patients in Placebo group had no data for week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Divaza | Placebo
Number analyzed (Participants) | 56 | 57
Participants | 56 | 51
Statistical Analysis 1: Comparison: Divaza vs Placebo; Test type: Superiority; p = 0.0272, Fisher Exact — A priori threshold for statistical significance is split evenly between primary and secondary endpoints. α=0.025

3. Other Pre Specified Outcome: Change in Mean Level of Preformed LP Products (Mainly Lipid Hydroperoxides).
Description: Based on laboratory evaluation. Change in mean level of preformed LP products, predominantly lipid hydroperoxides after 12-week therapy versus baseline.
  The following kinetic parameters of chemiluminescence were measured: rapid chemiluminescence flare amplitude reflecting the stationary level of lipid hydroperoxides.
Time Frame: 12 weeks of the observation period
Population: 1 patient in Divaza group had no laboratory data.
Measure: Mean (Standard Deviation); unit: Mcmol / L
Arm/Group | Divaza | Placebo
Number analyzed (Participants) | 63 | 59
Mcmol / L
  Level of preformed LPO products at baseline | 72.5 (14.1) | 72.8 (12.9)
  Level of preformed LPO products after 12 weeks | 67.7 (13.1) | 69.9 (11.7)
  ∆ between baseline and after 12 weeks | -3.2 (9.6) | -2.9 (8.0)
Statistical Analysis 1: Comparison: Divaza vs Placebo; This analysis applies to ∆ between baseline and after 12 weeks row; Test type: Superiority; p = 0.8762, t-test, 2 sided

4. Other Pre Specified Outcome: Change in Mean Value of Lipoprotein Ability for Oxidation.
Description: Based on laboratory evaluation. Change in mean value of lipoprotein ability for oxidation after 12-week therapy versus baseline.
  For plasma, draw blood into an EDTA tube and gently invert the tube 8 to 10 times to mix the anticoagulant. Centrifuge the tube, remove the stopper and draw off approximately 2/3 of the upper plasma layer into a labeled transfer tube using a transfer pipet bulb. Plasma must be separated from cells within 45 minutes of venipuncture. Measurement of oxidized LDL (oxLDL) has been incorporated into clinical practice in the diagnosis and treatment of lipid disorders (such as diabetes mellitus), atherosclerosis, and various liver and renal diseases, especially as it pertains to the evaluation of oxidative stress. Oxidized LDL-particles are considered to be an important driving factor in the pathophysiology of atherosclerosis and oxLDL measurement has been used to test the efficacy of CVD drugs (eg, statins) to reduce oxidative stress.
Time Frame: 12 weeks of the observation period.
Population: 1 patient in Divaza group had no laboratory data.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Divaza | Placebo
Number analyzed (Participants) | 63 | 59
mV
  LP ability for oxidation at baseline | 1027.3 (204.7) | 993.8 (264.1)
  LP ability for oxidation after 12 weeks | 1024.1 (226.7) | 1040.6 (217.7)
  ∆ between baseline and after 12 weeks | -12.1 (192.1) | 57.0 (241.5)
Statistical Analysis 1: Comparison: Divaza vs Placebo; This analysis applies to ∆ between baseline and after 12 weeks row; Test type: Superiority; p = 0.2082, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Change in Mean Value of NO Products Serum Concentration.
Description: Based on laboratory evaluation. Change in the mean concentration of nitrites and nitrates in serum after 12-week therapy versus baseline. Griess Reaction assay.
  In the Griess reaction, first reported by Johann Peter Griess in 1879 as a method of analysis of nitrite (NO2-), nitrite reacts under acidic conditions with sulfanilic acid (HO3SC6H4NH2) to form a diazonium cation (HO3SC6H4-Ntriple bondN+) which subsequently couples to the aromatic amine 1-naphthylamine (C10H7NH2) to produce a red-violet coloured (λmax ≈ 540 nm), water-soluble azo dye (HO3SC6H4-Ndouble bondN-C10H6NH2).
Time Frame: 12 weeks of the observation period.
Measure: Mean (Standard Deviation); unit: μmol per liter
Arm/Group | Divaza | Placebo
Number analyzed (Participants) | 7 | 8
μmol per liter
  NO-3 level at baseline | 41.3 (14.9) | 69.0 (28.9)
  NO-3 level (after cuff test) at baseline | 38.4 (16.5) | 79.1 (33.5)
  NO-3 level after 12 weeks | 51.7 (23.9) | 63.3 (36.8)
  NO-3 level (after cuff test) after 12 weeks | 64.0 (15.6) | 61.1 (27.9)
  NO-2 level at baseline | 35.9 (16.0) | 62.8 (28.0)
  NO-2 level (after cuff test) at baseline | 31.8 (16.1) | 69.6 (32.3)
  NO-2 level after 12 weeks | 43.9 (22.2) | 52.5 (35.9)
  NO-2 level (after cuff test) after 12 weeks | 57.0 (14.5) | 51.0 (25.9)
  NO level at baseline | 5.4 (2.3) | 6.3 (4.1)
  NO level (after cuff test) at baseline | 6.6 (1.8) | 9.5 (4.0)
  NO level after 12 | 7.8 (3.9) | 10.7 (4.5)
  NO level (after cuff test) after 12 weeks | 7.0 (2.8) | 10.1 (5.2)
Statistical Analysis 1: Comparison: Divaza vs Placebo; This analysis applies to NO-3 data; Test type: Superiority; p = 0.0038, Mixed Models Analysis — The p-value associated with "treatment*visit" interaction between Divaza and Placebo treatment groups. Model includes cuff test status, treatment, visit and treatment*visit interaction
Statistical Analysis 2: Comparison: Divaza vs Placebo; This analysis applies to NO-2 data; Test type: Superiority; p = 0.0018, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Divaza vs Placebo; This analysis applies to NO data; Test type: Superiority; p = 0.46, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

6. Other Pre Specified Outcome: Change in Mean Value of Platelet Aggregation.
Description: Based on laboratory evaluation. Change in mean platelet aggregation after 12-week therapy versus baseline.
Time Frame: 12 weeks of the observation period.
Population: ADP-AP - platelet aggregation (PA) induced by adenosine diphosphate (ADP) ADR-AP - platelet aggregation (PA) induced by adrenaline (ADR)
Measure: Mean (Standard Deviation); unit: percentage aggregation
Arm/Group | Divaza | Placebo
Number analyzed (Participants) | 7 | 8
percentage aggregation
  ADP-PA at baseline | 46.9 (13.8) | 44.6 (14.1)
  ADP-PA (after cuff test) at baseline | 45.0 (14.0) | 51.9 (15.7)
  ADP-PA after 12 weeks | 45.3 (12.5) | 46.3 (9.4)
  ADP-PA (after cuff test) after 12 weeks | 49.7 (14.6) | 52.5 (11.6)
  ADR-PA at baseline | 48.4 (12.2) | 47.8 (16.4)
  ADR-PA (after cuff test) at baseline | 44.7 (13.3) | 53.1 (16.8)
  ADR-PA after 12 weeks | 47.7 (11.8) | 51.4 (11.3)
  ADR-PA (after cuff test) after 12 weeks | 54.1 (8.6) | 57.4 (14.6)
Statistical Analysis 1: Comparison: Divaza vs Placebo; This analysis applies to ADP-PA data; Test type: Superiority; p = 0.88, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Divaza vs Placebo; This analysis applies to ADR-PA data; Test type: Superiority; p = 0.93, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: During the treatment period - 12 weeks (start after taking the first dose of the study drug, during the entire period of the study therapy and within 24 hours after the last dose of the study drug).
Arm/Group | Divaza | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/59
Other Adverse Events (participants affected / at risk) | 5/64 | 3/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Divaza (N=64) | Placebo (N=59)
Odinophagy (Gastrointestinal disorders) | 1 (1) | 0 (0) — Sore throat when swallowing
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Increased blood pressure (Investigations) | 0 (0) | 1 (1) — Increase in blood pressure to 235/120 mmHg
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Tick bite

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT03485495/Prot_SAP_000.pdf